CLINICAL TRIAL: NCT02230423
Title: Trigeminale Endonasale Perzeption, Ein Prädiktor für Das Outcome Einer Septumplastik - Eine Prospektive Kohortenstudie Mit Klinischen Und Biologischen Untersuchungen
Brief Title: Trigeminal Endonasal Perception: A Predictor for Septoplasty Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SM_31_01_2014; KEK-ZH-Nr: 2013-0545 (Other: Zurich Ethics Committee)
Record Dates: First submitted 2014-04-28; First posted 2014-09-03 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Empty Nose Syndrome
Keywords: Functional nasal surgery; Empty Nose Syndrome (ENS)
MeSH Terms: interventions — Nasal Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients receiving nose surgery (Experimental): Patients in need of nose surgery, before and after surgery; or only after successful surgery, then with or without "Empty Nose Syndrome".
  Interventions: Procedure: Nasal surgery

INTERVENTIONS:
Procedure: Nasal surgery
  Other Names: Septoplasty; Turbinoplasty; Removal of turbinates and septum parts

SUMMARY:
This study investigates wether patients with increased trigeminal perception threshold and low expression of TRP channels have more often nasal blockage despite functionally successful nasal surgery (TRP channel = transient receptor potential channel).

DETAILED DESCRIPTION:
The aim of this study is to find out wether patients with high trigeminal perception threshold (=decreased intranasal sensibility) and low expression of TRP channels of the mucosa suffer more often from impaired nasal breathing after surgery. This could lead to the identification of prognostic factors and therefore prevention of nasal surgery with bad outcome.

Further, differences between patients with empty nose syndrome and asymptomatic patients after extended intranasal surgery, concerning trigeminal perception and TRP channel expression will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary septoplasty and/or turbinoplasty
* Patients suffering from empty nose syndrome after measurably successful nasal surgery
* Patients with removed turbinates and/or septum, not suffering from ENS (i.e. tumor patients)

Exclusion Criteria:

* Patients with known neurologic disorders that could compromise perception threshold measurements
* Patients with known allergies/intolerance to test agents that are used to measure perception thresholds (Cineol=Eucalypt; Menthol, CO2= Carbon Dioxide)
* Inability to judge or understand the testing or the informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-05; Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Measurement of subjective nasal breathing impairment after surgery depending on trigeminal perception threshold and TRP channel expression | Up to 1 year post-surgery

SECONDARY OUTCOMES:
Differences between trigeminal perception threshold as as well as TRP expression levels in patients with postoperative empty nose syndrome and patients with subjectively unimpaired nasal breathing after extended intranasal surgery | Up to 1 year post-op

CONTACTS AND LOCATIONS:
Overall Officials: Michael Soyka, Dr.med., Principal Investigator — Zurich University Hospital
Locations (1):
- Zurich University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No